CLINICAL TRIAL: NCT00330499
Title: A Randomised Trial of Radical Chemo/Radiotherapy vs Radiotherapy Alone in the Definitive Management of Localised Muscle Invasive TCC of the Urinary Bladder
Brief Title: Efficacy Study of Adding Chemotherapy to Radiotherapy for Treating Bladder Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROG 02.03; NHMRC 243100
Record Dates: First submitted 2006-05-25; First posted 2006-05-26 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Transitional Cell Carcinoma of Urinary Bladder
Keywords: Locally invasive; Bladder cancer; Chemoradiotherapy; Efficacy; Organ conservation
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Synchronous chemo / radiation therapy
  Interventions: Drug: Cisplatin; Radiation: External beam radiation treatment
- B (Active Comparator): Radiation Alone
  Interventions: Radiation: External beam radiation treatment

INTERVENTIONS:
Drug: Cisplatin — Weekly Cisplatin 35mg/m2 x 6 doses, IV administration
  Other Names: Cisplatuin Ebewe, Cisplatin Injection
  Arms: A
Radiation: External beam radiation treatment — 64Gy reference dose in 32 fractions over 6.5 weeks
  Other Names: Radiation

SUMMARY:
The purpose of this study is to define the optimal management of localised transitional cell carcinoma (TCC) of the urinary bladder. The main objective is to evaluate whether chemoradiation is superior to radiotherapy alone.

DETAILED DESCRIPTION:
Whilst concurrent chemo-radiation is increasingly being looked upon as the treatment of choice for patients referred for bladder preservation, the study by the NCI of Canada (Coppin CM, Gospodarowicz MK et al.Improved Local Control of Invasive Bladder Cancer by Concurrent Cisplatin and Pre-operative or Definitive Radiation.J. of Clinical Oncol. 14(11): 2901-2907, 1996) is the only randomised trial to show some superiority of concurrent Cisplatin and radiation treatment over radiation alone in increasing pelvic tumour control. There was no impact on overall survival. However, this study had relatively small subject numbers and included two distinct treatment options. In one group the patients were treated with a bladder sparing approach and in the other by pre-operative therapy and cystectomy with the type of definitive treatment being decided upon by both the treating Specialist and patient. At 5 years the pelvic failure rates in the radiation alone and chemo-radiation arms were 59% and 40% respectively. With half of the patients in each group having had planned cystectomy as part of their treatment regimen, the above rates of local relapse (especially in the chemo-radiation arm) are disappointing.

Given the concerns with the above study, and the continuing paucity of randomised phase III studies comparing chemo-radiation with radiation alone, there lies an opportunity for Australasian centres to take up the challenge. For this study, the proposed schedule for the chemo-radiation arm is to be the same as that being investigated in our previous phase II study (six weekly doses of Cisplatin plus radiation to a dose of 64Gy in 32 fractions over 6.5 weeks). This will be compared with radical radiation alone (64Gy in 32 fractions over 6.5 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven TCC of the urinary bladder. Mixed tumours comprising predominantly TCC and elements of squamous or adenomatous metaplasia or carcinoma are also eligible.
* Clinically and radiologically localised T2, T3 or T4a non-bulky disease (<= 7cm in maximum dimension), N0, M0.

If radiological evaluation of a lymph node is interpreted as "positive" this must be evaluated further by either lymph node sampling or percutaneous needle biopsy. Patients with histologically confirmed lymph node metastases will not be eligible.

* Maximal TUR.

N.B. Previous:

1. partial cystectomy;
2. endoscopic resection of bladder tumour/s;
3. intravesical chemotherapy; or
4. intravesical BCG

does not exclude the patient from being eligible. However, the patient should have an adequate functioning bladder (this should be clarified with the referring Urologist and if need be voiding volumes should be measured).

* Creatinine clearance >= 50ml/minute by calculation or measurement.
* A white blood cell count >= 3.5 x 10^9/L with an absolute neutrophil count >= 1.5 x 10^9/L and a platelet count >= 100 x 10^9/L.
* ECOG status of 0, 1 or 2.
* No age limit applies provided the patient is mentally, physically and geographically capable of undergoing treatment and follow-up.
* No significant intercurrent morbidity.

Exclusion Criteria:

* Pure squamous carcinomas or adenocarcinomas.
* Extensive or multifocal CIS change in the bladder.
* T3 or T4a tumours unsuitable for curative treatment (i.e. > 7cm in any dimension), T4b, node positive and metastatic disease.
* Presence of ureteric obstruction due to tumour infiltration at the UO not amenable to stenting.
* Previous radiation treatment to the pelvis.
* Previous significant pelvic surgery.
* Significant bowel or gynaecological inflammatory disease.
* Creatinine clearance < 50ml/minute by calculation or measurement. A white blood cell count < 3.5 x 10^9/L with an absolute neutrophil count < 1.5 x 10^9L and/or a platelet count < 100 x 10^9/L.
* Other considerations making patient unfit for Cisplatin therapy.
* Prior or concurrent malignancy of any other site unless disease-free for greater than 5 years, except for:

  1. non-melanoma skin cancer, and/or
  2. (a) Stage T1 well differentiated prostatic carcinoma in men, and In situ carcinoma of the cervix in women.
* Bladder tumour - biopsy only. These patients must be referred back for more adequate resections or else should not be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2002-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Invasive local failure at 3 years | 3 years

SECONDARY OUTCOMES:
Complete response (CR) rate at 3 months from randomisation | 3 months
Disease-free survival | Final analysis when all patients have been followed for 3 years. (approx. 7 years from start of trial)
Overall survival | Final analysis when all patients have been followed for 3 years. (approx. 7 years from start of trial)
Cystectomy-free survival | Final analysis when all patients have been followed for 3 years. (approx. 7 years from start of trial)
Acute and late toxicity | Interim analyses will be performed on an annual basis.
Pattern of failure (local, regional, distant) | Final analysis when all patients have been followed for 3 years. (approx. 7 years from start of trial)
Quality of life measures | Final analysis when all patients have been followed for 3 years. (approx. 7 years from start of trial)

CONTACTS AND LOCATIONS:
Overall Officials: Kumar Gogna, Study Chair — Mater Centre - South Brisbane
Locations (22):
- Australia (17):
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Nepean Cancer Care Centre, Penrith, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - Mater Centre - South Brisbane, Brisbane, Queensland
  - Townsville Hospital, Douglas, Queensland
  - Royal Brisbane Hospital, Herston, Queensland
  - East Coast Cancer Centre, Tugun, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Andrew Love Cancer Care Centre, Geelong Hospital, Geelong, Victoria
  - Alfred Hospital, Prahran, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- New Zealand (5):
  - Auckland Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Palmerston North Hospital, Palmerston North
  - Wellington Hospital, Wellington

REFERENCES:
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au